CLINICAL TRIAL: NCT00676247
Title: Cerebral Blood Flow Parameters and Neurobehavioral Development in Full-Term Infants and Very Low Birth Weight Preterm Infants at Term Age
Brief Title: Cerebral Blood Flow Parameters and Neurobehavioral Development in Infants at Term Age
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Suh-Fang Jeng, National Taiwan University
Other Study IDs: 200802011R
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Premature Birth
Keywords: Ultrasonography; Doppler; Hemodynamics; Neurobehavioral development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- preterm: Very-low-birth-weight preterm infants with brain lesion
- full-term: Healthy fullterm infants

SUMMARY:
Although several studies have contrasted the hemodynamics of cerebral arteries using cranial Doppler ultrasound between full-term and preterm infants, the assessments were mostly conducted in the first days of life. Furthermore, the clinically significant hemodynamic parameter has been established from a small sample of infants that its validity on other populations remains unclear. Therefore, the purpose of this study is twofold:

1. to examine the hemodynamics of cerebral arteries in full-term and very low birth weight preterm infants at term age
2. to assess the validity of the hemodynamic parameters in relation to concurrent neurobehavioral function.

This study will enroll normal full-term infants and very low birth weight preterm infants who have no major neonatal disease. Cranial Doppler ultrasound examination will be performed on all infants at term age. Hemodynamic parameters will include peak systolic velocity, end diastolic velocity, resistance index and pulsatility index for the bilateral anterior cerebral arteries and middle cerebral arteries. Neurobehavioral development will be administered on the same day using the Neonatal Neurobehavioral Examination- Chinese version.

DETAILED DESCRIPTION:
We estimate the sample size of this study based on the cerebral blood flow velocity data of Kempley's study that showed 7.2 ± 3.5 and 10.7 ± 2.4 cm/s for the MCAs in 13 preterm and 8 full-term infants, respectively. As the power is set at 0.8 and the α level is at 0.05, at least 17 subjects were required for each group. This study will include 20 full-term and 20 VLBW preterm infants who are born at the National Taiwan University Hospital (NTUH) and the Mackay Memorial Hospital (MMH), Taipei, Taiwan. Written informed consent will be obtained from the parents before participation in this study.

Cranial Doppler ultrasound and the NNE-C examinations will be performed within 5 days after birth on full-term infants and at post-menstrual age (PMA) of 40 weeks (± 1 week) on preterm infants in the baby room. If the examination time occurs after hospital discharge, assessment will be conducted in the baby room at NTUH or in the ultrasound examination room at MMH. The examinations will be performed when the babies show stable vital signs in daily activities. The NNE-C examination will be administered one hour prior to feeding to minimize distress. The NNE-C examination will be performed immediately after the ultrasound assessment. The two examinations will be performed by different examiners who were blind to each other's results. During brain Doppler ultrasound examination, each infant will be placed on the back in a baby crib or an incubator with his/her head in midline. Infant's behavioral state will be kept in the behavioral state of 1 (quiet sleep), 2 (active sleep), or 3 (drowsy) on Brazelton's classification to eliminate the impact on cerebral blood flow velocity.

Hemodynamic parameters will include PSV, EDV, RI, and PI from bilateral ACAs and MCAs as obtained by the pulse wave color Doppler. The ACA will be approached through the anterior fontanel on the sagittal plane and its blood flow velocity will be determined at the proximal part. The MCA will be approached under the transverse plane by placing the transducer on the temporal bone below the zygomatic arch. The flow velocity measurements will be obtained by Fourier transform analysis from homogeneous blood flow wave patterns over at least 3 cardiac cycles with good clear signals. Those signals that show complete and similar waveforms in the adjacent cycles and have high magnitudes with visible margin recognized from the background noise will be selected. The RI and PI are the ratio between the different velocities with the formulas: RI = (PSV-EDV) / PSV, PI = (PSV-EDV) / mean velocity. The whole ultrasound examination will take about 10 minutes.

ELIGIBILITY:
Fullterm group

Inclusion Criteria:

* birth weight higher than 2,500 g
* appropriate for gestational age
* gestation age within 38 and 42 weeks

Exclusion Criteria:

* chromosomal or congenital abnormalities

Preterm group

Inclusion Criteria:

* birth weight less than 1,500 g
* gestational age less than 37 weeks
* admission at the hospitals within 7 days after birth

Exclusion Criteria:

* chromosomal or congenital abnormalities

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns in the primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow velocity | post-conceptional age=40 weeks

SECONDARY OUTCOMES:
Neonatal Neurobehavioral Examination | post-conceptional age=40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Doctor, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan